CLINICAL TRIAL: NCT03289975
Title: Early Identification of Patients in Surgical Intensive Care With a Risk of Acute Respiratory Distress Following Visceral Surgery: Prognostic Value of Pulmonary Extravascular Water Revealed by Pulmonary Ultrasound.
Brief Title: Early Identification of Patients in Surgical Intensive Care With a Risk of Acute Respiratory Distress Following Visceral Surgery
Acronym: ODR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DRANSART BOUHEMAD 2016
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Digestive Surgery; Urinary Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pulmonary ultrasound — Collect the aeration profile for each lung quadrant: profile A, profile B1, profile B2, profile C. Calculate the aeration score from O to 36 (LUS (Lung ultrasound) score).

SUMMARY:
Today there are few studies in the literature involving patients in an ICU following major visceral surgery. There are thus few results about the prognostic value of pulmonary extravascular water in this population of patients, but also the prognostic value of pulmonary extravascular water measured at the bedside using pulmonary ultrasound.

In addition, pulmonary ultrasound will be combined with echocardiography to measure left ventricular function (LVEF) and to study the profile of the mitral valve to assess filling pressure in patients with immediate post-operative ventilation. This will make it possible to distinguish between increases in pulmonary extravascular water associated with high filling pressure and increased pulmonary water associated with low filling pressure: characteristic of lesional oedema.

The aim of this study is to determine the prognostic value of extravascular pulmonary water (PEVW) diagnosed using pulmonary ultrasound in patients admitted to an ICU following scheduled or emergency visceral surgery in the onset of acute respiratory distress requiring invasive mechanical ventilation, or prolonged post-operative intubation, or non-invasive.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing scheduled or emergency visceral surgery and admitted to an ICU following the intervention.

Exclusion Criteria:

* Chest surgery
* ASA (American Society of Anesthesiologists) 4 or more
* Refusal of the patient
* Pregnant women
* Spontaneously-breathing patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing digestive or urinary surgery and requiring post-operative intensive care
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Onset of post-operative acute respiratory distress | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Dransart-Raye O, Roldi E, Zieleskiewicz L, Guinot PG, Mojoli F, Mongodi S, Bouhemad B. Lung ultrasound for early diagnosis of postoperative need for ventilatory support: a prospective observational study. Anaesthesia. 2020 Feb;75(2):202-209. doi: 10.1111/anae.14859. Epub 2019 Sep 23. PMID 31549404